CLINICAL TRIAL: NCT03138174
Title: OneTouch Verio Flex System Accuracy Evaluation
Acronym: OTVFSA
Status: Completed | Type: Observational
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Other Study IDs: WI3052203
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus
Keywords: Blood Glucose Monitor System Accuracy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: None Retained — Capillary blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Diabetes: One group consisting of diabetic subjects
  Interventions: Device: OneTouch Verio Flex Blood Glucose Monitoring System

INTERVENTIONS:
Device: OneTouch Verio Flex Blood Glucose Monitoring System — Blood Glucose Monitoring System

SUMMARY:
Clinical System Accuracy Evaluation of the CE Marked One Touch Verio Flex blood glucose monitoring device as per requirements stated in ISO 15197:2015. To meet the requirements, glucose samples must be distributed over the operating range of the blood glucose monitor as stipulated in ISO:15197

DETAILED DESCRIPTION:
Clinical System Accuracy Evaluation of the CE Marked One Touch Verio Flex blood glucose monitoring device as per requirements stated in ISO 15197:2015.

ELIGIBILITY:
Summary of Inclusion Criteria:

* All Subjects must be registered into the LFSS Patient Registry to participate in the study.
* Each Participant must read and sign the approved Informed Consent Form.
* Diabetes Diagnosis - Participants should be diagnosed with some form of diabetes for system accuracy.

Summary of Exclusion Criteria:

> Subjects not enrolled in the LFSS Patient Registry are not eligible to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of subjects diagnosed with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
To meet the requirements of ISO 15197:2015 | Four weeks
  In order to meet the requirements of ISO 15197:2015
  1. For each lot individually, 95% of the individual glucose results shall fall within either +0.83 mmol/L (+ 15 mg/dL) of the average measured values of the reference measurement procedure at glucose concentration intervals < 5.55 mmol/L (< 100 mg/dL) or within + 15 % at glucose concentrations > 5.55 mmol/L (> 100 mg/dL).
  2. 99% of individual glucose measured values shall fall within zones A and B of the Consensus Error Grid for type 1 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Patrick, Principal Investigator — National Health Service, United Kingdom
Locations (3):
- United Kingdom (3):
  - Diabetes Centre, Birmingham Heartlands Hospital, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Highland Diabetes Institute, Inverness

IPD SHARING:
Plan to Share IPD: No
De identified data may be shared by way of study reports and publications